CLINICAL TRIAL: NCT06124846
Title: Determining the Effect of Six Weeks of Cannabis Abstinence on Fronto- Striatal fMRI Markers in Adolescents With Cannabis Use Disorder (ABSCAN)
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: PSYCH-2023-32396
Record Dates: First submitted 2023-11-03; First posted 2023-11-09 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Cannabis Use Disorder

STUDY DESIGN:
Intervention Model Description: This parallel intervention study will collect fMRI data in adolescents ages 15-18 years old with and without CUD at three different timepoints over the course of their intervention. abstinence. Age- and sex-matched adolescents with no lifetime history of cannabis use will also complete the protocol.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- control (No Intervention): Age- and sex-matched adolescents with no lifetime history of cannabis use will also complete the protocol.
- CB-Abst (Experimental): adolescents ages 15-18 years old with CUD use randomized to CB-Abst
  Interventions: Behavioral: CB-Abst
- CB-MON (Experimental): adolescents ages 15-18 years old with CUD use randomized to CB-Mon
  Interventions: Behavioral: CB-Mon

INTERVENTIONS:
Behavioral: CB-Abst — incentivized, biochemically verified abstinence via contingency management
  Arms: CB-Abst
Behavioral: CB-Mon — monitoring with no required abstinence
  Arms: CB-MON

SUMMARY:
The goal of this study is to understand the changes in neural correlates of reward in adolescents with and without Cannabis Use Disorder (CUD). The study will collect functional magnetic resonance imaging (fMRI) data at 3 different timepoints with the primary goals of understanding striatal reward-based activation during a Monetary Incentive Delay Task and fronto-striatal fMRI resting-state functional connectivity. The study will also explore self-reported impulsivity. The long-term goal is to advance scientific understanding of neural changes associated with cannabis abstinence and inter-individual variability that cannot be otherwise measured in preexisting observational cohorts such as the Adolescent Brain Cognitive Development Study.

This parallel intervention study will collect fMRI data in adolescents ages 15-18 years old with and without CUD at three different timepoints over the course of their intervention. Utilizing a validated paradigm, adolescents with CUD will be randomized to 6-weeks of either incentivized, biochemically verified abstinence via contingency management or monitoring with no required abstinence. Age- and sex-matched adolescents with no lifetime history of cannabis use will also complete the protocol. Participants will complete 8 study visits (3 with fMRI scans) involving urinalysis to confirm cannabis self-report and measures of impulsivity. Participants may additionally and optionally (1) complete daily remote self-report assessments of cannabis use, impulsivity, and mood throughout the 6-week treatment period, and (2) continue participation for an additional 6-week monitoring period after the treatment period, during which they complete daily remote self-report assessments of cannabis use, impulsivity, and mood.

ELIGIBILITY:
Inclusion Criteria:

* Male and female adolescents between the ages of 15 and 18 (inclusive).
* Have a parent or legal guardian who is able and willing to provide written informed consent.
* Competent and willing to provide written informed assent (participants <18) or consent (participants=18).
* Native English speaker.
* Have a parent or legal guardian who is fluent in English.
* Able to commit to 8 study visits in approximately 60 days (6 weeks).
* Able to safely participate in the protocol and appropriate for outpatient level of care, in the opinion of the PI.
* No active psychosis or current use of antipsychotic medications.
* Participants taking psychotropic medications will be included if the medications have been stable for 6 weeks and are expected to remain stable for the duration of their study participation (i.e., through the third MRI).
* For CB-Abst (n=24) and CB-Mon (n=20) groups: at least 5 days of use per week on average in the past two months and meet DSM-V cannabis use disorder (CUD; at least Mild) criteria. Cannabis use reported within seven days of baseline visit. Positive qualitative urine toxicology test at baseline for THC. No immediate plan to discontinue cannabis use.
* For Con (n=20): no lifetime history of cannabis use. Negative qualitative urine toxicology test at baseline for THC. No immediate plans to begin cannabis use.
* For optional components (A: daily remote assessments during and/or (B) after treatment period): access to a personal device (e.g., smartphone or computer) on which to complete daily remote assessments.

Exclusion Criteria:

* Past twelve-month history of substance use disorders (except for Cannabis Use Disorder in CB-Abst and CB-Mon), assessed via semi-structured psychodiagnostics interview at baseline.
* Current daily nicotine use (e.g., via electronic and/or combustible cigarettes).
* Contraindications for MRI (ascertained via participant and parent report), including but not limited to:

  1. Metal implants such as surgical clips or pacemakers, or history of working with metal, unless the possibility of a metal fragment can be ruled out by recent orbital scans.
  2. Prior head trauma with neurological sequelae.
  3. Claustrophobia.
  4. Weight incompatible with MRI safety.
  5. Pregnancy.
* Previous or current diagnosis of psychosis, cognitive disability, or bipolar disorder.
* Active suicidality.
* Taking a psychotropic medication that has not reached stability criterion (same medication type and dose for 6 weeks with no planned changes over the study period).
* Any other medical or psychiatric condition deemed serious or contraindicated for any study procedures by Dr. Tervo-Clemmens.

Ages: 15 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 64 (Estimated)
Dates: Start 2024-04-01 (Actual); Primary Completion 2028-04-15 (Estimated); Study Completion 2028-04-15 (Estimated)

PRIMARY OUTCOMES:
Brain activation during Monetary Incentive Delay Task (reward processing) | baseline, week3, week 6
  A neural measure of reward activation will be defined as the difference between reward positive vs negative feedback in the standardized Harvard Oxford Striatal atlas during the MID Task.
Brain connectivity during resting-state functional neuroimaging protocol | baseline, week 3, week 6
  A neural measure of reward-circuitry connectivity will be defined as the correlation values between standardized striatal and salience and orbitofrontal and salience cortical networks

SECONDARY OUTCOMES:
Self-reported Impulsivity via UPPS-P scale | baseline, weeks 1,2,3,4,5 and 6
  Self-reported impulsivity will be defined by Total and Premeditation (lack of), Urgency, Sensation Seeking, Perseverance (lack of) scores

CONTACTS AND LOCATIONS:
Overall Officials: Brenden Tervo-Clemmens, PhD, Principal Investigator — University of Minnesota
Locations (1):
- University of Minnesota, Minneapolis, Minnesota, United States